CLINICAL TRIAL: NCT03416998
Title: Effect Of Pre-Game Photobiomodulation On Muscle Recovery In Professional Soccer Players: Randomized, Cross-Over, Sham-Controlled, Triple-Blind, Clinical Trial
Brief Title: Photobiomodulation On Muscle Recovery In Professional Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Daniela Ap. Biasotto-Gonzalez, Doctor, University of Nove de Julho
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PHOTOBIOMODULATION
Record Dates: First submitted 2017-11-26; First posted 2018-01-31 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Muscle Development
Keywords: Photherapy; Photobiomodulation; Creatine Kinase; Soccer; Muscle Recovery
MeSH Terms: interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phototherapy Active (Active Comparator): Phototherapy active group will be administered 30 minutes prior to the soccer match as well as 48 h after the match in direct contact with the skin with light pressure at predetermined sites: nine on the knee extensor muscles, six on the knee flexor muscles and two on the gastrocnemius muscle on both lower limbs.
  Interventions: Other: phototherapy
- Placebo Phototherapy (Placebo Comparator): Phototherapy placebo group will be administered 30 minutes prior to the soccer match as well as 48 h after the match in direct contact with the skin with light pressure at predetermined sites: nine on the knee extensor muscles, six on the knee flexor muscles and two on the gastrocnemius muscle on both lower limbs.
  For placebo treatment, the same procedures and treatment times will be employed, but the equipment will be set in placebo mode. Only the researcher in charge of programming the device will have knowledge regarding which treatment is being used. However, the programmer will not participate in the execution of the treatment, evaluations or data analysis
  Interventions: Other: phototherapy

INTERVENTIONS:
Other: phototherapy — Phototherapy will be performed using clusters of 12 diodes (Table 1); four 905 nm diodes (mean power of 0.3125 mW and peak power of 12.5 W for each diode; 250 Hz), four 875 nm diodes (mean power of 17.5 mW for each diode) and four 640 nm diodes (mean power of 15 mW for each diode). The device manufactured by Multi Radiance Medical® (Solon, OH, USA) will be used due to its high quality, ample use in clinical practice and due to the fact that no national companies manufacture diode clusters with the characteristics required for the proposed project.

SUMMARY:
Background: Photobiomodulation with low-level laser therapy (LLLT) has been widely used in clinical practice for diverse purposes, such as modulation of the inflammatory process, acceleration of the tissue repair process, pain relief and the enhancement of post-exercise recovery. Studies have demonstrated a beneficial interaction between photobiomodulation and the production of creatine kinase, with a reduction in the release of this marker of muscle damage when laser and/or LEDs is administered prior to high-intensity physical activity. The aim of the proposed study is to determine the influence of pre-exercise phototherapy on post-exercise muscle recovery.

Methods: A randomized, cross-over, sham-controlled, double-blind, clinical trial is proposed. The participants will be healthy professional soccer players aged 15 to 20 years from the same team with a body mass index within the ideal range (20 to 25 kg/m2) and no history of lower limb musculoskeletal injuries or surgery or back surgery in the previous six months. The athletes will be allocated to two groups based on the previously calculated sample size and will be blinded to allocation. Creatine kinase will be measured and the subjective perception of fatigue will be determined for each participant. The volunteers will then be randomly allocated to Group A, which will receive active phototherapy, and Group B, which will receive sham phototherapy. The athletes will undergo reevaluations immediately after as well as 48 hours after a football match. The data will be submitted to statistical analysis and the level of significance will be set to 5%.

ELIGIBILITY:
Inclusion Criteria:

* Healthy professional soccer players aged 15 to 20 years from the same team with a body mass index in the ideal range (20 to 25 kg/m2) will be included in the study.

Exclusion Criteria:

* A history of musculoskeletal injuries and/or surgeries in the lower limbs or back surgery in the previous six months

Ages: 15 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2018-02-10 (Actual)

PRIMARY OUTCOMES:
Muscle recovery | 30 Minutes
  Analysis of creatine kinase

SECONDARY OUTCOMES:
Subjective muscle recovery | 30 Minutes
  Analysis of subjective fatigue scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nove de Julho, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No